CLINICAL TRIAL: NCT00612404
Title: Symptoms and Endoscopic Results in Consideration of Pretreatment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Kai Richter, AstraZeneca Germany
Other Study IDs: 1312004008
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Gastrointestinal Diseases
Keywords: gastrointestinal disorder; endoscopy; patient with gastrointestinal disorders for whom an endoscopy is performed and who is treated with esomeprazole afterwards.
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with gastrointestinal disorders who need an endoscopy.

SUMMARY:
Under daily routine conditions and without any intervention by the sponsor regarding the selection of subjects, diagnostic procedures, therapeutic decisions (medicinal and non- medicinal therapy, dose, duration, etc.), routine assessments, the participating physicians (i.e. gastroenterologists) are asked to document relevant data in patients with gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastrointestinal disorders who need an endoscopy.

Exclusion Criteria:

* limitiations; possible risks; warnings; contraindications mentioned in the SPC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: gastroenterologists; specialists
Sampling Method: Probability Sample
Enrollment: 16255 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
to gain insight into the relationship between subjective gastrointestinal symptoms and findings of a laryngopharyngeal-esophagogastric endoscopy with respect to the medicinal pre-therapy;

SECONDARY OUTCOMES:
to gain insight into the currently used treatment strategies with esomeprazole depending on endoscopic findings.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Richter, MD, Study Chair — Medical Department AstraZeneca Germany